CLINICAL TRIAL: NCT04165369
Title: Observational Study to Evaluate the Epidemiology of Surgical-induced Acute Kidney Injury
Acronym: Epis-AKI
Status: Completed | Type: Observational
Sponsor: University Hospital Muenster (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 01-AnIt-19
Record Dates: First submitted 2019-10-30; First posted 2019-11-18 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Acute Kidney Injury (AKI)
Keywords: Acute kidney injury; injury; surgery
MeSH Terms: conditions — Acute Kidney Injury; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with extended surgical exposures: Patients with extended surgical exposures requiring postoperative observation.

SUMMARY:
The evaluation of an accurate occurrence rate for AKI is of great importance for health policy, quality initiatives as well as for designing clinical trials.

The primary objective is to prospectively evaluate the incidence of AKI within 72 h after extended surgical procedures that require admission to an observation unit.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is a severe clinical complication with increasing incidence and is associated with adverse short- and long-term outcomes resulting in a major health care burden worldwide. The introduction of consensus classification systems has enhanced the awareness for AKI. The evaluation of an accurate occurrence rate for AKI is of great importance for health policy, quality initiatives as well as for designing clinical trials. However, analyzing AKI from existing databases is often limited by missing data elements, especially the inclusion of the urine output criteria. Missing data and the use of different definitions before the consensus classification are the reasons for large variations in reported occurrences of surgical induced AKI.

The primary objective is to prospectively evaluate the incidence of AKI within 72 h after extended surgical procedures that require admission to an observation unit (e.g., Intensive Care Unit, Intermediate Care, Post Anesthesia Care Unit) using the latest consensus definition for AKI (Kidney Disease: Improving Global Outcomes criteria) and a standardized data collection instrument and to assess the dependence of AKI on preoperative and intraoperative factors.

Method: International prospective, observational, multi-center, cross-sectional cohort study

Eligible patients will be identified during preoperative assessment. All eligible patients will be approached to obtain written consent.

ELIGIBILITY:
Inclusion Criteria:

* major elective or emergency surgery procedures with a duration of at least 2 h
* admission to the intensive care unit, intermediate care unit after surgery informed consent

Exclusion Criteria:

* preexisting acute kidney injury
* acute kidney injury within the last 3 months
* end stage renal disease with dialysis dependency
* kidney transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing extended surgical procedure and the need for postoperative observation
Sampling Method: Probability Sample
Enrollment: 10568 (Actual)
Dates: Start 2020-06-09 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Incidence of Acute Kidney Injury | 72 hours after extended surgery
  Occurrence of acute kidney injury according to the Kidney Disease: Improving Global Outcomes (KDIGO) criteria

SECONDARY OUTCOMES:
Severity of acute kidney injury (number of patients with KDIGO stage 1, KDIGO stage 2 or KDIGO stage 3) | 72 hours after extended surgery
  Definition and classification of acute injury according to the KDIGO (Kidney Disease: Improving Global Outcomes) clinical practice guidelines on acute kidney injury
Number of patients with renal replacement therapy | up to 90 days after extended surgery
Mortality | up to 90 days after extended surgery
Hospital stay | up to 90 days after extended surgery (until discharge)
Intensive Care Unit stay | up to 90 days after extended surgery (until discharge)
Major Adverse Kidney Events (MAKE) | up to 90 days after extended surgery
  combined endpoint consisting of mortality, renal replacement therapy, persistent renal dysfunction defined as serum-creatinine >= 1.5 times as compared to baseline serum-creatinine

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Zarbock, MD, PhD, Study Chair — University Hospital Muenster, Dept. of Anesthesiology, Intensive Care and Pain Medicine
Locations (82):
- University of Alabama, Birmingham, Alabama, United States
- Egypt (3):
  - Mansoura University Hospitals, Al Mansurah
  - Alexandria University, Alexandria
  - Tanta University Faculty of Medicine, Tanta
- France (17):
  - CHU d'Angers, Angers
  - Centre Hospitalier Simone Veil de Blois, Blois
  - CHU de Bordeaux, Bordeaux
  - Centre de Lutte contre le Cancer Francois Baclesse, Caen
  - Hopital Privé Sévigné, Cesson-Sévigné
  - Hopital Huriez - CHU de Lille, Lille
  - Clinique Chénieux, Limoges
  - Hopital Edouard Herriot, Lyon
  - Centre Hospitalier des Pays de Morlaix, Morlaix
  - CHU de Nices, Nice
  - Hopital Bichat, Paris
  - Hopital Maison Blance, Reims
  - Clinique Sainte-Anne, Strasbourg
  - CHG Tarbes, Tarbes
  - Clinique Pasteur Toulouse, Toulouse
  - Hopital Robert Schuman-Groupe UNEOS, Vantoux
  - Gustave Roussy, Villejuif
- Germany (5):
  - Kliniken Maria Hilf, Mönchengladbach
  - Herz Jesu Krankenhaus Münster Hiltrup, Münster
  - University Hospital Muenster, Münster
  - St. Josef-Stift Sendenhorst, Sendenhorst
  - Universitätsklinikum Tübingen, Tübingen
- Italy (4):
  - Ospedale di Montebelluna, Montebelluna
  - University of Palermo, Palermo
  - Cardioanestesia - Azienda Ospedaliera San Carlo di Potenza, Potenza
  - Ospedale Sant'Eugenio di Roma, Rome
- Libya (2):
  - National Heart Center Tripoli, Tripoli
  - Tripoli Central Hospital, Tripoli
- Mater Dei Hospital, Birkirkara, Malta
- University Clinic, Skopje, North Macedonia
- Palestinian Territories (2):
  - Al-Shifa Medical Complex, Gaza
  - Alia Governmental Hospital, Hebron
- Russia (3):
  - Kemerovo Cardiology Centre, Kemerovo
  - Bakulev Scientific Center for Cardiovascular Surgery, Moscow
  - Polenov Neurosurgical Institute, Saint Petersburg
- Almana General Hospital, Khobar, Saudi Arabia
- Slovenia (2):
  - University Medical Centre Maribor, Ljubljana
  - Splosna bolnisnica Murska Sobota, Murska Sobota
- Spain (11):
  - Hospital Universitario Araba, Alava
  - Hospital Universitario Funcacion Alcorcón, Alcorcón
  - Urology Fundación Puigvert, Barcelona
  - Donostia University Hospital, Donostia / San Sebastian
  - Hospital Cliínico Universitario Virgen de las Nieves, Granada
  - Hospital Universitario de Gran Canaria Doctor Negrin, Las Palmas de Gran Canaria
  - San Pedro Hospital, Logroño
  - Hospital Ramón y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Infanta Leonor University Hospital, Madrid
  - Son Llatzer University Hospital, Palma de Mallorca
- Turkey (Türkiye) (29):
  - Cukurova University, Adana
  - Akdeniz University Hospital, Akdeniz
  - Ankara City Hospital, Ankara
  - Ibn Sina Hospital, Ankara
  - Kahramanmaras Sutcu Imam University, Ankara
  - Balikesir University, Balıkesir
  - Uludag University, Bursa
  - University of Health Sciences, Bursa
  - Health Sciences University Medical School, Derince
  - Düzce University, Düzce
  - Gazi University Hospital, Gazi
  - Acibadem MAA Ünv. Altunizade Ä'Acibadem, Istanbul
  - Acibadem MAA Ünv. Atakent Acibadem, Istanbul
  - Haseki Egitim Arastirma, Istanbul
  - Istanbul University - Cerrahpasa, Istanbul
  - Istanbul University, Istanbul
  - Koc University Hospital, Istanbul
  - Prof. Dr. Cemil Tascioglu City Hospital, Istanbul
  - Yeditepe, Istanbul
  - Dokuz Eylül Üniversitesi, Izmir
  - Izmir Democracy University School of Medicine, Izmir
  - Health Sciences University Kartal, Kartal
  - Inönü University Hospital, Malatya
  - Manisa, Medical Faculty, Manisa
  - Suleyman Demirel University School of Medicine, Merkez
  - Mersin University, Mersin
  - Mayis University, Samsun
  - Karadeniz Technical University, Trabzon
  - University Faculty of Medicine, Trakya

REFERENCES:
- [Derived] Meersch M, Weiss R, Strauss C, Albert F, Booke H, Forni L, Pittet JF, Kellum JA, Rosner M, Mehta R, Bellomo R, Rosenberger P, Zarbock A; EPIS-AKI Investigators. Acute kidney disease beyond day 7 after major surgery: a secondary analysis of the EPIS-AKI trial. Intensive Care Med. 2024 Feb;50(2):247-257. doi: 10.1007/s00134-023-07314-2. Epub 2024 Jan 29. PMID 38285051
- [Derived] Zarbock A, Weiss R, Albert F, Rutledge K, Kellum JA, Bellomo R, Grigoryev E, Candela-Toha AM, Demir ZA, Legros V, Rosenberger P, Galan Menendez P, Garcia Alvarez M, Peng K, Leger M, Khalel W, Orhan-Sungur M, Meersch M; EPIS-AKI Investigators. Epidemiology of surgery associated acute kidney injury (EPIS-AKI): a prospective international observational multi-center clinical study. Intensive Care Med. 2023 Dec;49(12):1441-1455. doi: 10.1007/s00134-023-07169-7. Epub 2023 Jul 28. PMID 37505258
- [Derived] Weiss R, Saadat-Gilani K, Kerschke L, Wempe C, Meersch M, Zarbock A; EPIS-AKI Investigators. EPIdemiology of Surgery-Associated Acute Kidney Injury (EPIS-AKI): study protocol for a multicentre, observational trial. BMJ Open. 2021 Dec 30;11(12):e055705. doi: 10.1136/bmjopen-2021-055705. PMID 35588372

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-07-16): https://cdn.clinicaltrials.gov/large-docs/69/NCT04165369/SAP_000.pdf